CLINICAL TRIAL: NCT06980714
Title: Efficacy of Powered Versus Manual Toothbrushes on Full-Mouth Bleeding and Plaque Scores in Patients With Stage 3 or 4 Periodontitis
Brief Title: Powered vs. Manual Toothbrushing in Stage 3-4 Periodontitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Davide Pietropaoli, PI Davide Pietropaoli, Professor, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Verb n. 25 del 14/09/22 Addend
Record Dates: First submitted 2025-05-08; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis; Dental Plaque; Gingival Bleeding
Keywords: Periodontitis; Full-Mouth Plaque Score; Full-Mouth Bleeding Score; Home Oral Hygiene
MeSH Terms: conditions — Periodontitis; Dental Plaque; Gingival Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to either a powered toothbrush group or a manual toothbrush group. Each group follows the same oral hygiene protocol, with standardized brushing instructions. The two groups are followed in parallel over a 6-month period without crossover.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinical investigator who interacts with participants and the outcomes assessor responsible for evaluating clinical indices (FMBS and FMPS) are both blinded to group allocation. Participants are instructed not to disclose the type of toothbrush they are using. The masking helps ensure unbiased data collection and outcome assessment throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual (Active Comparator): Participants assigned to this arm use a manual toothbrush (TePe Select Soft) to perform twice-daily toothbrushing for at least 2 minutes. Brushing technique and duration are standardized through individual instruction at baseline. Participants are instructed not to use any additional oral hygiene aids, including mouthwash or interdental cleaners. Brushing sessions are monitored and recorded via a smartphone app to ensure compliance with the 2-minute minimum duration.
  Interventions: Behavioral: Manual
- Powered (Experimental): Participants assigned to this arm use a powered toothbrush (Oral-B iO6) to perform twice-daily toothbrushing for at least two minutes. Brushing technique and duration are standardized through individual instruction at baseline. Participants are instructed not to use any additional oral hygiene aids, including mouthwash or interdental cleaners. The powered toothbrush provides consistent brushing performance, and participants are monitored to ensure compliance with the 2-minute minimum duration.
  Interventions: Behavioral: Powered

INTERVENTIONS:
Behavioral: Powered — The intervention involves the use of the Oral-B iO6 powered toothbrush, which provides oscillating-rotating brushing action with personalized feedback via its smart pressure sensor and app integration. Participants in this group are instructed to brush for at least two minutes twice daily. The toothbrush is designed to ensure consistent brushing performance, with real-time feedback on brushing technique and duration, allowing for improved oral hygiene habits. The intervention aims to standardize brushing duration and technique, eliminating potential variations found with manual brushing.
  Arms: Powered
Behavioral: Manual — The intervention involves the use of the TePe Select Soft manual toothbrush, which features soft bristles for gentle yet effective plaque removal. Participants in this group are instructed to brush for at least two minutes twice daily, with guidance on proper brushing technique. To ensure compliance with the brushing duration, participants are required to use a smartphone app that tracks and records their brushing sessions. The manual toothbrush allows for participant control over brushing pressure and technique, with no additional oral hygiene aids allowed during the study period.
  Arms: Manual

SUMMARY:
This study compares the effectiveness of powered and manual toothbrushes in reducing gum bleeding and dental plaque in people with stage 3 or 4 periodontitis. All participants are trained to brush for at least two minutes twice a day. The goal is to find out whether using a powered toothbrush leads to better oral hygiene results than a manual one, when brushing time is standardized. The study will measure bleeding and plaque levels at the beginning and over a 6-month period.

DETAILED DESCRIPTION:
This single-blind, randomized controlled trial evaluates the clinical effectiveness of powered versus manual toothbrushing in patients newly diagnosed with stage 3 or 4 periodontitis. Participants are randomly assigned to one of two groups: powered toothbrush (Oral-B iO6) or manual toothbrush (TePe Select Soft). All participants receive standardized oral hygiene instructions and are instructed to brush twice daily for a minimum of two minutes. Manual brush users are required to use a smartphone app to monitor and record brushing duration. The use of adjunctive oral hygiene aids, such as mouthwash or interdental cleaners, is restricted throughout the study period. The primary clinical outcomes are full-mouth bleeding score (FMBS) and full-mouth plaque score (FMPS), measured at baseline and at follow-ups of 7 days, 1 month, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* Diagnosis of stage 3 or 4 periodontitis based on clinical and radiographic examination
* Retaining at least 16 natural teeth
* Ability to follow oral hygiene instructions and compliance with the study protocol
* Willingness to refrain from using additional oral hygiene products (e.g., mouthwash, interdental cleaners) during the study
* Ability to provide informed consent

Exclusion Criteria:

* Presence of systemic conditions that may affect oral health (e.g., uncontrolled diabetes, immunocompromised states)
* Pregnancy or breastfeeding
* Ongoing use of antibiotics or other medications that could interfere with gum health
* Severe dental conditions (e.g., tooth mobility > 2, advanced root resorption)
* Prior use of a powered toothbrush within the last 6 months
* Participation in another clinical trial that could interfere with study outcomes
* Inability or unwillingness to comply with study requirements or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Full-Mouth Bleeding Score (FMBS) | FMBS will be assessed at baseline and at 7 days, 1 month, 3 months, and 6 months following the intervention.
  The Full-Mouth Bleeding Score (FMBS) will be used to assess the level of gingival bleeding upon gentle probing across all teeth in the mouth. This measure will evaluate the overall gum health of participants and will help compare the effectiveness of the powered versus manual toothbrushes in reducing gingival inflammation. FMBS will be recorded at baseline, 7 days, 1 month, 3 months, and 6 months to monitor changes in bleeding over time.

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure (SBP and DBP) | SBP and DBP will be measured at baseline, 1 month, 3 months, and 6 months.
  Systolic and Diastolic Blood Pressure (SBP and DBP) will be measured using the Omron M6 device, following the European Society of Hypertension (ESH) guidelines for proper measurement techniques. Blood pressure will be recorded to evaluate any potential changes related to the oral hygiene interventions. Measurements will be taken at baseline, 1 month, 3 months, and 6 months to monitor any trends in blood pressure variation over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Pietropaoli, DDS, PhD, Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: Yes
Yes, individual participant data (IPD) will be shared with qualified researchers upon request, following ethical guidelines and the necessary approvals. The data will be anonymized and shared through a secure data repository to ensure privacy and confidentiality.
Time Frame: Starting 12 months after publication; available for 3 years
Access Criteria: Researchers with a methodologically sound proposal and ethics approval